CLINICAL TRIAL: NCT04838028
Title: Mesh and Fixation Combinations in Laparoendoscopic Groin Hernia Repair: Association With Chronic Postoperative Pain. A Swedish Hernia Registry Study.
Brief Title: Chronic Postoperative Pain After Laparoendoscopic Groin Hernia Repair
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other); Swedish Hernia Registry (Unknown)
Responsible Party: Principal Investigator, Bengt Novik, MD, PhD, SSOD, Karolinska Institutet
Other Study IDs: Bengan IV
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain; Chronic Pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — tetraethylpyrazine; tetra-4-amidinophenoxypropane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (9):
- Standard polypropylene mesh: Density > 50 g/square meter
  Interventions: Procedure: TEP; Procedure: TAPP; Procedure: Other or unspecified laparoendoscopic groin hernia repair
- Lightweight mesh: * A mesh based on either polypropylene or polyester. Some variants contain purely 1 polymer. Others are composite, ie, contain also an absorbable material.
  * The density < 50 g/square meter (when applicable, after partial absorption).
  * In this study, the property of light weight will trump the material, ie, any lightweight mesh having been registered as, eg, "Polyester mesh", will be reclassified as "Lightweight mesh".
  Interventions: Procedure: TEP; Procedure: TAPP; Procedure: Other or unspecified laparoendoscopic groin hernia repair
- Fixation with metal tacks: Non-absorbable metal staples or tacks
  Interventions: Procedure: TEP; Procedure: TAPP; Procedure: Other or unspecified laparoendoscopic groin hernia repair
- Fixation with absorbable tacks: Absorbable synthetic staples or tacks
  Interventions: Procedure: TEP; Procedure: TAPP; Procedure: Other or unspecified laparoendoscopic groin hernia repair
- Fibrin glue fixation: Biologic glue/sealant produced from human donor blood
  Interventions: Procedure: TEP; Procedure: TAPP; Procedure: Other or unspecified laparoendoscopic groin hernia repair
- Non-fixation: Mesh is deployed without fixation
  Interventions: Procedure: TEP; Procedure: TAPP; Procedure: Other or unspecified laparoendoscopic groin hernia repair
- 3D mesh: A polypropylene mesh with a preformed anatomic shape corresponding to the inner preperitoneal curvature of the groin.
  The category does not differentiate between standard and lightweight variants.
  Interventions: Procedure: TEP; Procedure: TAPP; Procedure: Other or unspecified laparoendoscopic groin hernia repair
- Progrip fixation: Absorbable (Velcro type of) microhooks. The particular meshes come with prefabricated Progrip microhooks. Progrip = Registered trademark.
  Interventions: Procedure: TEP; Procedure: TAPP; Procedure: Other or unspecified laparoendoscopic groin hernia repair
- Polyester mesh: Polyester-based mesh. This category does not differentiate between standard and lightweight variants. If a mesh was initially registered under this category by the surgeon, but identified being a lightweight mesh by the researchers, it will be re-classified as "Lightweight mesh".
  Interventions: Procedure: TEP; Procedure: TAPP; Procedure: Other or unspecified laparoendoscopic groin hernia repair

INTERVENTIONS:
Procedure: TEP — Laparoendoscopic totally extraperitoneal mesh repair of groin hernia
Procedure: TAPP — Laparoscopic transabdominal mesh repair of groin hernia
Procedure: Other or unspecified laparoendoscopic groin hernia repair — "Other" refers to any laparoendoscopic mesh repair specified as not being either TEP or TAPP, eg, "intraperitoneal onlay mesh" (IPOM).

SUMMARY:
The study attempts to quantify the relative risks for chronic postoperative inguinal pain (CPIP) depending on different combinations of mesh and mesh fixation. For this purpose the investigators will analyze data from the Swedish Hernia Registry (SHR).

DETAILED DESCRIPTION:
This is an open cohort study design where the investigators will analyze existing data that have been prospectively collected in the Swedish Hernia Registry (SHR), which covers > 95% of all groin hernia repairs in Sweden. The very large cohort of approximately 25,000 primary TEP (totally extraperitoneal) and TAPP (transabdominal preperitoneal) repairs enable assessment of the relative risks for CPIP depending on different combinations of mesh and mesh fixation. Each participant was entered at the date of surgery when demographic and intraoperative data were registered. The possible presence of CPIP after 1 year postoperative was evaluated with a PROM questionnaire.

ELIGIBILITY:
Inclusion Criteria:

All laparoendoscopic repairs for groin hernia that have been registered in the SHR from September 1, 2012, until December 31, 2018.

Exclusion Criteria:

* Open repairs.
* Hernioplasties that were converted from laparoscopic to open surgery.
* Bilateral repairs.
* Surgery merely for hernia (eg obturator) other than lateral, medial or femoral.
* Age < 15 years.
* Patients not having a 10-digit state-assigned Patient Identification Number.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An unselected, consecutive nationwide cohort during 7 years, with a 1-year follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 15360 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Relative risk for postoperative pain at 1 year | 1 year
  Chronic postoperative inguinal pain, measured by the Short Form Inguinal Pain Questionnaire (sf-IPQ)

SECONDARY OUTCOMES:
Reoperation | 1-8 years
  Reoperation due to recurrence, during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Novik, MD, Principal Investigator — Dept of Clinical Sciences, Karolinska Institutet, Danderyd Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No
The dataset analyzed in the current study was retrieved from the Swedish Hernia Registry. It is not publicly available and cannot be requested from the authors.
  To access the data, a separate application must be made to the Registry.

REFERENCES:
- [Background] Novik B, Nordin P, Skullman S, Dalenback J, Enochsson L. More recurrences after hernia mesh fixation with short-term absorbable sutures: A registry study of 82 015 Lichtenstein repairs. Arch Surg. 2011 Jan;146(1):12-7. doi: 10.1001/archsurg.2010.302. PMID 21242440
- [Background] Novik B, Hagedorn S, Mork UB, Dahlin K, Skullman S, Dalenback J. Fibrin glue for securing the mesh in laparoscopic totally extraperitoneal inguinal hernia repair: a study with a 40-month prospective follow-up period. Surg Endosc. 2006 Mar;20(3):462-7. doi: 10.1007/s00464-005-0391-3. Epub 2006 Jan 19. PMID 16424986
- [Background] Franneby U, Gunnarsson U, Andersson M, Heuman R, Nordin P, Nyren O, Sandblom G. Validation of an Inguinal Pain Questionnaire for assessment of chronic pain after groin hernia repair. Br J Surg. 2008 Apr;95(4):488-93. doi: 10.1002/bjs.6014. PMID 18161900
- [Background] Olsson A, Sandblom G, Franneby U, Sonden A, Gunnarsson U, Dahlstrand U. The Short-Form Inguinal Pain Questionnaire (sf-IPQ): An Instrument for Rating Groin Pain After Inguinal Hernia Surgery in Daily Clinical Practice. World J Surg. 2019 Mar;43(3):806-811. doi: 10.1007/s00268-018-4863-8. PMID 30478683
- [Background] Novik B, Sandblom G, Ansorge C, Thorell A. Association of Mesh and Fixation Options with Reoperation Risk after Laparoscopic Groin Hernia Surgery: A Swedish Hernia Registry Study of 25,190 Totally Extraperitoneal and Transabdominal Preperitoneal Repairs. J Am Coll Surg. 2022 Mar 1;234(3):311-325. doi: 10.1097/XCS.0000000000000060. PMID 35213495